CLINICAL TRIAL: NCT06701084
Title: Molecular Genetic Mechanisms of Infantile Epilepsies and the Impact of Genetic Diagnosis: Gene-Shortening Time of Evaluation in Pediatric Epilepsy Services (Gene-STEPS)
Brief Title: Molecular Genetic Mechanisms of Infantile Epilepsies and the Impact of Genetic Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alissa D'Gama, Instructor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1K23NS140397 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Epilepsy; Infantile Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genomic Sequencing (Experimental): All enrolled infants receive the intervention (genomic sequencing, including rapid genome sequencing). Comprehensive genomic analyses will be performed to identify genetic diagnoses. Genetic results will be returned to families and infants will be followed until 2.5 years old to evaluate the impact of genetic diagnosis using quantitative validated outcome measures and qualitative parent interviews.
  Interventions: Genetic: Genomic Sequencing

INTERVENTIONS:
Genetic: Genomic Sequencing — Genomic sequencing data will be comprehensively analyzed for pathogenic variants that explain the participants epilepsy.

SUMMARY:
The goal of this study is to discover new genetic causes of infantile epilepsies and evaluate the impact of these discoveries on infants with epilepsy and their families.

DETAILED DESCRIPTION:
Infantile epilepsies are common, affecting 1 in 1000 infants, and are associated with significant morbidity, mortality, healthcare costs, and caregiver burden. Although most infantile epilepsies are believed to have genetic causes, most infants with epilepsy remain genetically "unsolved" and the full genetic landscape of infantile epilepsies is unknown, which limits our ability to develop precision therapies and ultimately improve outcomes for this vulnerable population. This study aims to discover new genetic causes of infantile epilepsies and evaluate the impact of these discoveries on infants with epilepsy and their families, contributing to knowledge that will inform our scientific understanding of normal and abnormal brain development and guide clinical care and implementation of precision medicine for infants with epilepsy.

ELIGIBILITY:
Infant Criteria

Inclusion Criteria:

* Seizure onset at less than 12 months of age
* Enrollment within 6 weeks of seizure-related presentation
* Patient at Boston Children's Hospital

Exclusion Criteria:

* Simple febrile seizures
* Acute provoked seizures (e.g., due to sepsis, hemorrhage, electrolyte abnormality, cerebral infarction, hypoxic ischemic encephalopathy, non-accidental injury)
* Genetic or acquired cause of epilepsy already identified, including brain magnetic resonance imaging findings consistent with a specific genetic etiology (e.g., tuberous sclerosis complex)
* Deceased prior to enrollment

Parent Criteria Inclusion Criteria - Parent of eligible infant (see above)

Exclusion Criteria

- Not the legal guardian of the eligible infant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | Collected after return of genetic results approximately 2 weeks after infant is enrolled
  The diagnostic yield of genomic sequencing will be calculated as the percentage of enrolled infants with epilepsy who receive a genetic diagnosis.
Short-term clinical utility of genetic testing | Collected after return of genetic results approximately 2 weeks after infant is enrolled
  The short-term clinical utility of genetic testing will be evaluated using the validated C-GUIDE measure. The C-GUIDE total score will be compared between infants with epilepsy who did vs did not receive a genetic diagnosis.
Parent-perceived (personal) utility of genetic testing | Collected when infant is 2.5 years old
  The parent-perceived utility of genetic testing will be evaluated using the validated GENE-U measure. The GENE-U total score will be compared between infants with epilepsy who did vs did not receive a genetic diagnosis.

SECONDARY OUTCOMES:
Developmental progress | Collected when infant is 2.5 years old
  Developmental progress will be evaluated using the Bayley Scales of Infant and Toddler Development Fourth Edition. The cognitive, language, and motor subscale scores will be compared between infants with epilepsy who did vs did not receive a genetic diagnosis.
Seizure frequency | Collected at return of genetic results approximately 2 weeks after infant is enrolled and when infant is 2.5 years old
  The seizure frequency will be evaluated using the seizure frequency outcome measure developed by the American Academy of Neurology and dichotomized as decrease vs no decrease between the two timepoints. The percentage of infants with this outcome will be compared between infants with epilepsy who did vs did not receive a genetic diagnosis.
Parental experiences with genetic testing | Collected when infant is 2.5 years old
  This outcome will be evaluated using a qualitative approach. Semi-structured interviews will be performed with a subset of parents using purposive sampling and will be analyzed using a grounded theory iterative approach.

CONTACTS AND LOCATIONS:
Overall Officials: Alissa M D'Gama, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States